CLINICAL TRIAL: NCT04298931
Title: Fluid Responsiveness Prediction Using Pulse Pressure Variation - Integrating Ventilator Settings
Brief Title: Prediction of the Effect of Fluid Administration Using Arterial Pressure and Ventilator Data During Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-245-19
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-04

CONDITIONS: Hypovolemia; Fluid Overload
MeSH Terms: conditions — Hypovolemia; Edema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing open abdominal surgery
  Interventions: Other: Series of ventilator settings

INTERVENTIONS:
Other: Series of ventilator settings — Before a planned fluid administration, the investigators will apply a series of 10 ventilator settings for 30 seconds each.
  The settings are the following combinations of respiratory rate (RR) and tidal volume (TV):
  RR (min^-1), TV (ml/kg predicted body weight)
  31, 6
  31, 8
  24, 6
  24, 8
  17, 6
  17, 8
  10, 4
  10, 6
  10, 8
  10, 10
  (the order of the respiratory rates: 17 to 31, will be randomized. 10/min will always be last. Tidal volume is always applied from lowest to highest for each respiratory rate).

SUMMARY:
It is well known, that patients with circulatory impairment sometimes, but not always, benefit from intravenous fluids. Predicting if a fluid administration will improve circulation is therefore of substantial clinical interest.

Ventilator treatment induces cyclic variation in blood pressure due to interaction between the lungs and the heart. This variation is minor, but its amplitude may be used for guiding fluid administration.

However, this method of using ventilator-induced variation in blood pressure to predict the effect of fluid administration was developed when different settings for ventilator treatment was recommended, compared with today. With today's recommend ventilator treatment, the method is, unfortunately, less reliable.

The investigators will investigate how different ventilator settings influence variation in blood pressure, and the investigators will test if this knowledge allows us to better predict the effect of a fluid administration, by taking the ventilator settings into account.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled open abdominal surgery.
* Scheduled treatment with Aarhus University Hospital's goal-directed therapy protocol (hemodynamic monitoring).

Exclusion Criteria:

* Left ventricular ejection fraction ≤ 40 %
* Irregular heart rhythm (e.g. atrial fibrillation or frequent ectopic beats)
* Known right ventricular dysfunction (if reported qualitatively in pre-operative assessment or objectively via Tricuspid Annular Plane Systolic Excursion (TAPSE) < 17 mm)
* Pregnancy
* Prior participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at department of abdominal surgery, Aarhus University Hospital, scheduled for open abdominal surgery with planned use of Aarhus University Hospital's goal-directed therapy protocol (hemodynamic monitoring).
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
>10% Increase in stroke volume from before to after a fluid bolus. (Fluid responsiveness) | From two minutes before to two minutes after a fluid administration.
  A patient is considered a fluid responder if they have a >10% increase in stroke volume (pulse contour analysis by the Edwards EV1000 with a FloTrac sensor).
  Pre-fluid stroke volume is calculated as the median stroke volume estimate in the two minutes immediately preceding the fluid bolus.
  Post-fluid stroke volume is calculated as the median stroke volume estimate in the two minutes immediately following the fluid bolus.
  Change in stroke volume is calculated as: 100% * (Post-fluid stroke volume - Pre-fluid stroke volume) / Pre-fluid stroke volume

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Enevoldsen J, Brandsborg B, Juhl-Olsen P, Rees SE, Thaysen HV, Scheeren TWL, Vistisen ST. The effects of respiratory rate and tidal volume on pulse pressure variation in healthy lungs-a generalized additive model approach may help overcome limitations. J Clin Monit Comput. 2024 Feb;38(1):57-67. doi: 10.1007/s10877-023-01090-6. Epub 2023 Nov 16. PMID 37968547